CLINICAL TRIAL: NCT03338855
Title: DAPAMAAST: A Double-blind, Randomized, Phase IV, Mechanistic, Placebo-controlled, Cross-over, Single-center Study to Evaluate the Effects of 5 Weeks Dapagliflozin Treatment on Insulin Sensitivity in Skeletal Muscle in Type 2 Diabetes Mellitus Patients.
Brief Title: Effects of 5 Weeks Treatment With Dapagliflozin in Type 2 Diabetes Patients on How the Hormone Insulin Acts on Sugar Uptake in Muscles.
Acronym: DAPAMAAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D1690C00047; 2016-003991-27 (EudraCT Number)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2; Skeletal Muscle Insulin Sensitivity
Keywords: T2DM, insulin resistance, skeletal muscle, mitochondria, dapagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Active Comparator): Patients will receive dapagliflozin 10 mg in tablet for a maximum of 40 days based on randomization sequence in Period 1.
  Patients that received 10 mg dapagliflozin in the first treatment period will receive matching placebo in the second treatment period for a maximum of 40 days.
  Interventions: Drug: Dapagliflozin
- Placebo matching to dapagliflozin (Placebo Comparator): Patients will receive matching placebo in tablet for a maximum of 40 days based on randomization sequence.
  Patients who received placebo in the first treatment will receive 10 mg dapagliflozin in the second treatment period, for a maximum of 40 days
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — The study consist of 5 weeks treatment period 1, 6-8 weeks wash-out period and 5 weeks treatment period 2.
  The patient will be administered dapagliflozin 10 mg during Period 1 or Period 2.

SUMMARY:
The purpose of this study is to investigate the effects of 5 weeks treatment with dapagliflozin in type 2 diabetes patients on how the hormone insulin acts on sugar uptake in muscles.

DETAILED DESCRIPTION:
To investigate if dapagliflozin improves skeletal muscle insulin sensitivity expressed as corrected glucose disposal rate (cGDR) in comparison with placebo after 5-week double blind treatment. Insulin sensitivity will be determined using a 2-step euglycemic hyperinsulinemic clamp (EHC) procedure

ELIGIBILITY:
Inclusion Critieria:

1. Patients are able to provide signed and dated written informed consent prior to any study specific procedures.
2. Women are post-menopausal (defined as at least 1 year post cessation of menses) and aged ≥ 45 and ≤ 70 years. Males are aged ≥ 40 years and ≤ 70 years. Patients should have suitable veins for cannulation or repeated venipuncture.
3. Patients are diagnosed with T2DM for at least the last 6 months.
4. Patients are on no other anti-diabetic drug treatment, or on stable maximum 3000 mg daily dose metformin treatment and/or on stable dose of a DPPIV inhibitor treatment for at least the last 3 months5. HbA1c levels ≥6.0% (=42 mmol/mol) and ≤9.0% (75 mmol/mol).
5. Have a body mass index (BMI) ≤ 35 kg/m2.

Exclusion Criteria:

1. Involvement in the planning and conduct of the study (applies to both AstraZeneca staff and staff at third party vendor or at the investigational sites).
2. Previous enrolment in the present study or participation in another clinical study with an investigational product during the last 3 months or as judged by the Investigator.
3. History of or presence of any clinically significant disease or disorder including a recent (< 3 months) cardiovascular event which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study or influence the results or the patient's ability to participate in the study.
4. Clinical diagnosis of Type 1 diabetes, maturity onset diabetes of the young, secondary diabetes or diabetes insipidus.
5. Unstable/rapidly progressing renal disease or estimated Glomerular Filtration Rate < 60 mL/min (Cockcroft-Gault formula).
6. Clinically significant out of range values of serum levels of either alanine aminotransferase (ALT), aspartate aminotransferase (AST) or alkaline phosphatase (ALP) in the Investigator's opinion.
7. Contraindications to dapagliflozin according to the local label.
8. Use of antidiabetic drugs other than metformin within 3 months prior to screening.
9. Weight gain or loss > 5 kg in the last 3 months, ongoing weight-loss diet (hypocaloric diet) or use of weight loss agents.
10. History of drug abuse or alcohol abuse in the past 12 months.
11. Any clinically significant abnormalities in clinical chemistry, hematology or urinalysis or other condition the Investigator believes would interfere with the patient's ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the patient at undue risk.
12. Plasma donation within one month of screening or any blood donation/blood loss > 500 mL within 3 months prior to screening or during the study.
13. Anemia defined as Hemoglobin (Hb) < 115 g/L (7.1 mM) in women and < 120 g/L (7.5 mM) in men.
14. Use of anti-coagulant treatment such as heparin, warfarin, platelet inhibitors, thrombin and factor X inhibitors.
15. Use of medication such as oral glucocorticoids, anti-estrogens or other medications that are known to markedly influence insulin sensitivity.
16. Use of loop diuretics.
17. Regular smoking and other regular nicotine use.
18. Any contra-indication to magnetic resonance imaging scanning. These contra-indications include patients with following devices:

    * Central nervous system aneurysm clip
    * Implanted neural stimulator
    * Implanted cardiac pacemaker of defibrillator
    * Cochlear implant
    * Metal containing corpora aliena in the eye or brain.
19. Patients, who do not want to be informed about unexpected medical findings, or do not wish that their physician be informed about coincidental findings, cannot participate in the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Maastricht, Netherlands

REFERENCES:
- [Derived] Op den Kamp YJM, Gemmink A, de Ligt M, Dautzenberg B, Kornips E, Jorgensen JA, Schaart G, Esterline R, Pava DA, Hoeks J, Schrauwen-Hinderling VB, Kersten S, Havekes B, Koves TR, Muoio DM, Hesselink MKC, Oscarsson J, Phielix E, Schrauwen P. Effects of SGLT2 inhibitor dapagliflozin in patients with type 2 diabetes on skeletal muscle cellular metabolism. Mol Metab. 2022 Dec;66:101620. doi: 10.1016/j.molmet.2022.101620. Epub 2022 Oct 21. PMID 36280113
- [Derived] Op den Kamp YJM, de Ligt M, Dautzenberg B, Kornips E, Esterline R, Hesselink MKC, Hoeks J, Schrauwen-Hinderling VB, Havekes B, Oscarsson J, Phielix E, Schrauwen P. Effects of the SGLT2 Inhibitor Dapagliflozin on Energy Metabolism in Patients With Type 2 Diabetes: A Randomized, Double-Blind Crossover Trial. Diabetes Care. 2021 Jun;44(6):1334-1343. doi: 10.2337/dc20-2887. Epub 2021 Apr 15. PMID 33858855
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690C00047&attachmentIdentifier=75766274-37ca-4c65-bd0b-5d8450cc900b&fileName=D1690C00047_CSP_redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1690C00047&attachmentIdentifier=ecc6c77d-916b-4286-acd2-5456fab108a6&fileName=D1690C00047_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double-blind, randomized, placebo-controlled, cross-over Phase IV mechanistic study which was conducted in 1 study center in the Netherlands between 05 March 2018 and 04 November 2019.
Pre-assignment Details: Eligible patients with Type 2 diabetes mellitus were randomized to a specific double-blind treatment sequence (either dapagliflozin then placebo or placebo then dapagliflozin). Each of the 2 treatment periods had a maximum duration of 40 days, separated by a wash-out period of 6 to 8 weeks.
Groups:
- Dapagliflozin 10 mg Then Placebo: Patients received an oral dose of 10 milligrams (mg) dapagliflozin, once daily for 5 weeks. After a wash-out period of 6 to 8 weeks, matched placebo tablets were taken orally, once daily for 5 weeks.
- Placebo Then Dapagliflozin 10 mg: Patients received placebo tablets (matched to dapagliflozin) taken orally, once daily for 5 weeks. After a wash-out period of 6 to 8 weeks, patients received an oral dose of 10 mg dapagliflozin, once daily for 5 weeks.
Period: Overall Study
Arm/Group | Dapagliflozin 10 mg Then Placebo | Placebo Then Dapagliflozin 10 mg
Started | 12 | 14
Received Treatment in Period 1 | 12 | 14
Received Treatment in Period 2 | 11 | 14
Completed | 11 | 14
Not Completed | 1 | 0
Not completed — Withdrawn as birth control pill stopped | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized analysis set consisted of all randomized patients.
Groups:
- Dapagliflozin 10 mg Then Placebo: Patients received an oral dose of 10 mg dapagliflozin, once daily for 5 weeks. After a wash-out period of 6 to 8 weeks, matched placebo tablets were taken orally, once daily for 5 weeks.
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10 mg Then Placebo | Placebo Then Dapagliflozin 10 mg | Total
Number analyzed (Participants) | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (4.7) | 64.4 (4.7) | 63.8 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 7 | 13 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 14 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Corrected Glucose Disposal Rate (cGDR) Measured as Change in Rate of Disposal (Delta RD) Basal vs High Insulin After 5 Weeks of Treatment
Description: Skeletal muscle insulin sensitivity was measured as cGDR (referred to as delta RD [basal vs high insulin]) using a 2-step 5.5 hour euglycemic hyperinsulinemic clamp (EHC) procedure in combination with infusion of D-glucose (6,6-D2) glucose. Delta RD (basal vs high insulin) was corrected for urinary glucose excretion and measured at the end of Treatment Periods 1 and 2.
Time Frame: At end (Week 5) of Treatment Periods 1 and 2
Population: The evaluable analysis set (clamp) was a subset of the randomized analysis set, consisting of patients who received at least 1 dose of any investigational product. Any patients with important procedure specific protocol deviations regarding the clamp method were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: micromole/kilogram body weight/minute
Groups:
- Dapagliflozin 10 mg: Patients received an oral dose of 10 mg dapagliflozin, once daily for 5 weeks in either Treatment Period 1 or Treatment Period 2.
- Placebo: Patients received an oral dose of placebo, once daily for 5 weeks in either Treatment Period 1 or Treatment Period 2.
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 22 | 22
micromole/kilogram body weight/minute | 8.523 [5.566 to 11.481] | 9.592 [6.634 to 12.549]
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Comparison of delta RD (basal vs high insulin) between dapagliflozin and placebo after 5 weeks of treatment was performed using a random effects analysis of variance model; Test type: Superiority; p = 0.3047, Linear Mixed Effects Model; A linear mixed model with treatment group, treatment sequence, and period as fixed effects and patient as random effect; Least Square (LS) Mean Difference = -1.068, 95% CI 2-sided [-3.183 to 1.047], Standard Error of Mean 1.014

2. Other Pre Specified Outcome: Change in Endogenous Glucose Production (EGP) After 5 Weeks of Treatment
Description: A 2-step 5.5 hour EHC in combination with infusion of 6,6-D2 glucose was used to determine rates of EGP at the end of Treatment Periods 1 and 2. Results of the change in EGP are presented as delta EGP (basal vs low insulin and basal vs high insulin).
Time Frame: At end (Week 5) of Treatment Periods 1 and 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: micromole/kilogram body weight/minute
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 22 | 22
micromole/kilogram body weight/minute
  Delta EGP (basal vs low insulin) | -4.656 [-5.494 to -3.817] | -2.591 [-3.790 to -2.112]
  Delta EGP (basal vs high insulin) | -10.803 [-11.726 to -9.880] | -8.512 [-9.435 to -7.589]
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Comparison of delta EGP (basal vs low insulin) between dapagliflozin and placebo after 5 weeks of treatment was performed using a random effects analysis of variance model; Test type: Superiority; p = 0.0036, Linear Mixed Effects Model; A linear mixed model with treatment group, treatment sequence, and period as fixed effects and patient as random effect; LS Mean Difference = -1.705, 95% CI 2-sided [-2.784 to -0.625], Standard Error of Mean 0.517
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; Comparison of delta EGP (basal vs high insulin) between dapagliflozin and placebo after 5 weeks of treatment was performed using a random effects analysis of variance model; Test type: Superiority; p < 0.0001, Linear Mixed Effects Model; A linear mixed model with treatment group, treatment sequence, and period as fixed effects and patient as random effect; LS Mean Difference = -2.292, 95% CI 2-sided [-3.146 to -1.438], Standard Error of Mean 0.409

3. Other Pre Specified Outcome: Change in Respiratory Exchange Ratio (RER) From Fasted State to Insulin Stimulated State After 5 Weeks of Treatment
Description: During the indirect calorimetry of the EHC test, respiratory gas exchange was measured using open air circuit respirometry with an automated ventilated hood system. Metabolic flexibility was determined by the change in RER from fasted state to insulin stimulated state at the end of Treatment Periods 1 and 2 and results are presented as delta RER (basal vs high insulin).
Time Frame: At end (Week 5) of Treatment Periods 1 and 2
Population: The evaluable analysis set (indirect calorimetry) was a subset of the randomized analysis set, consisting of patients who received at least 1 dose of any investigational product. Any patients with important procedure specific protocol deviations regarding the indirect calorimetry method were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 21 | 21
ratio | 0.101 [0.080 to 0.122] | 0.089 [0.068 to 0.110]
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Comparison of delta RER (basal vs high insulin) between dapagliflozin and placebo after 5 weeks of treatment was performed using a random effects analysis of variance model; Test type: Superiority; p = 0.1842, Linear Mixed Effects Model; A linear mixed model with treatment group, treatment sequence, and period as fixed effects and patient as random effect; LS Mean Difference = 0.012, 95% CI 2-sided [-0.006 to 0.030], Standard Error of Mean 0.009

4. Other Pre Specified Outcome: 24-Hour RER After 5 Weeks of Treatment
Description: RER was measured before and after meals over a 24-hour period.
Time Frame: At end (Week 5) of Treatment Periods 1 and 2
Population: The evaluable analysis set (chamber) was a subset of the randomized analysis set, consisting of patients who received at least 1 dose of any investigational product. Any patients with important procedure specific protocol deviations regarding the chamber method were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 24 | 24
ratio | 0.812 [0.803 to 0.821] | 0.835 [0.826 to 0.844]
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Comparison of 24-hour RER between dapagliflozin and placebo after 5 weeks of treatment was performed using a random effects analysis of variance model; Test type: Superiority; p = 0.0001, Linear Mixed Effects Model; A linear mixed model with treatment group, treatment sequence, and period as fixed effects and patient as random effect; LS Mean Difference = -0.023, 95% CI 2-sided [-0.033 to -0.013], Standard Error of Mean 0.005

5. Other Pre Specified Outcome: 24-Hour Energy Expenditure After 5 Weeks of Treatment
Description: Whole body energy expenditure was measured over a 24-hour period.
Time Frame: At end (Week 5) of Treatment Periods 1 and 2
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: megajoules/day
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 24 | 24
megajoules/day | 9.519 [9.017 to 10.020] | 9.628 [9.126 to 10.130]
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Comparison of energy expenditure between dapagliflozin and placebo after 5 weeks of treatment was performed using a random effects analysis of variance model; Test type: Superiority; p = 0.1095, Linear Mixed Effects Model; A linear mixed model with treatment group, treatment sequence, and period as fixed effects and patient as random effect; LS Mean Difference = -0.109, 95% CI 2-sided [-0.245 to 0.027], Standard Error of Mean 0.065

6. Other Pre Specified Outcome: Body Composition (Fat Mass and Lean Mass) After 5 Weeks of Treatment
Description: On Day 6, 7 or 8 of the end of treatment visit in both treatment periods, a Dual-energy X-ray absorptiometry (DEXA) scan was used to determine body composition.
Time Frame: At end (Week 5) of Treatment Periods 1 and 2
Population: The evaluable analysis set (DEXA) was a subset of the randomized analysis set, consisting of patients who received at least 1 dose of any investigational product. Any patients with procedure specific protocol deviations regarding the DEXA method were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: grams
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 24 | 24
grams
  Fat Mass | 25318.3 [22978.4 to 27658.1] | 25564.9 [23225.0 to 27904.8]
  Lean Mass | 59929.0 [56762.1 to 63095.8] | 60595.4 [57428.5 to 63762.3]
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Comparison of fat mass between dapagliflozin and placebo after 5 weeks of treatment was performed using a random effects analysis of variance model; Test type: Superiority; p = 0.6005, Linear Mixed Effects Model; LS Mean Difference = -246.7, 95% CI 2-sided [-1209.5 to 716.2], Standard Error of Mean 464.3 — A linear mixed model with treatment group, treatment sequence, and period as fixed effects and patient as random effect
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; Comparison of lean mass between dapagliflozin and placebo after 5 weeks of treatment was performed using a random effects analysis of variance model; Test type: Superiority; p = 0.0376, Linear Mixed Effects Model; A linear mixed model with treatment group, treatment sequence, and period as fixed effects and patient as random effect; LS Mean Difference = -666.5, 95% CI 2-sided [-1291.0 to -41.9], Standard Error of Mean 301.1

7. Other Pre Specified Outcome: Body Composition (Total Mass) After 5 Weeks of Treatment
Description: On Day 6, 7 or 8 of the end of treatment visit in both treatment periods a DEXA scan was used to determine body composition.
Time Frame: At end (Week 5) of Treatment Periods 1 and 2
Population: The evaluable analysis set (DEXA) was a subset of the randomized analysis set, consisting of patients who received at least 1 dose of any investigational product. Any patients with important procedure specific protocol deviations regarding the DEXA method were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 24 | 24
kilograms | 85.248 [81.608 to 88.888] | 86.504 [82.864 to 90.143]
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Comparison of total mass between dapagliflozin and placebo after 5 weeks of treatment was performed using a random effects analysis of variance model; Test type: Superiority; p = 0.0003, Linear Mixed Effects Model; LS Mean Difference = -1.256, 95% CI 2-sided [-1.854 to -0.657], Standard Error of Mean 0.289 — A linear mixed model with treatment group, treatment sequence, and period as fixed effects and patient as random effect

8. Other Pre Specified Outcome: Fibroblast Growth Factor 21 (FGF21) Area Under the Curve (AUC) in Plasma After 5 Weeks of Treatment
Description: From the end of Day 1 until the morning of Day 3 of the end of each treatment visit, the patients stayed in the metabolic chamber (36 hours). During this stay FGF21 was measured in plasma before and after meals and before bed-time to determine the AUC (last 24 hours).
Time Frame: At end (Week 5) of Treatment Periods 1 and 2
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: nanograms/liter/hour
Arm/Group | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 21 | 21
nanograms/liter/hour | 3310.415 [2626.919 to 3993.911] | 3554.716 [2871.270 to 4238.212]
Statistical Analysis 1: Comparison: Dapagliflozin 10 mg vs Placebo; Comparison of FGF21 AUC between dapagliflozin and placebo after 5 weeks of treatment was performed using a random effects analysis of variance model; Test type: Superiority; p = 0.1555, Linear Mixed Effects Model; LS Mean Difference = -244.301, 95% CI 2-sided [-590.002 to 101.401], Standard Error of Mean 165.168 — A linear mixed model with treatment group, treatment sequence, and period as fixed effects and patient as random effect

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported throughout the treatment period and including the follow-up period. Overall time frame up to a maximum of 19 weeks (including both 5-week treatment periods, 6-8 weeks wash-out and 5-10 days safety follow-up after last dose of study drug).
Description: In this study, collection of AE data was limited to the collection of serious AEs, discontinuation of investigational product due to an AE and potential diabetic ketoacidosis events only. The safety analysis set consisted of all patients who received at least 1 dose of study drug, with patients being analyzed and presented by treatment received, rather than as randomized.
Groups:
- Dapagliflozin 10mg: Patients received an oral dose of 10mg dapagliflozin, once daily for 5 weeks in either Treatment Period 1 or Treatment Period 2.
Arm/Group | Dapagliflozin 10mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT03338855/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03338855/SAP_001.pdf